CLINICAL TRIAL: NCT05845086
Title: The Effect of Multimedia-based Preoperative Patient Education Reinforced With Teach-back Method on Early Ambulation in Gynecological Surgery: a Randomized Controlled Trial
Brief Title: The Effect of Preoperative Patient Education on Early Ambulation in Gynecological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Ezgi Arslan, Principal Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Postoperative ambulation
Record Dates: First submitted 2023-04-12; First posted 2023-05-06 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Gynecologic Nursing; Surgery; Nurse's Role
Keywords: Early ambulation; Preoperative patient education; Nursing; Gynecologic surgery; Postoperative nursing care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Preoperative patient education) (Experimental): In addition to the usual care provided by the nurses, the intervention group will be provided with multimedia-supported written and verbal pre-operative patient training, reinforced by the teach-back method, created according to the literature.
  Interventions: Behavioral: Preoperative patient education
- Control group (Usual care) (No Intervention): The control group continued to receive the usual care

INTERVENTIONS:
Behavioral: Preoperative patient education — In this study, preoperative patient education will be given, reinforced with multimedia supported written and verbal teach-back method, created according to the literature. Videos of exercises used to increase postoperative mobilization (deep breathing exercise, coughing exercise, intensive spirometer use, etc.) will be taken by the researcher in a professional studio. The captured videos will be embedded in the PowerPoint presentation and presented to the patient with a tablet computer. The powerpoit presentation should be a maximum of 30 slides and the patient education should take a maximum of 30 minutes. Patients will be evaluated face-to-face on the 1st, 2nd, 3rd days after surgery and by phone on the 15th day. The prepared powerpoint presentation will be left with the patient as a printout. The prepared video will be given to the patient after the training with a program (via WhatsApp, e-mail, bluetooh) on their phones in accordance with the preferences of the patients.
  Arms: Intervention group (Preoperative patient education)

SUMMARY:
This study was planned as a randomized controlled study to test the effect of multimedia supported patient education reinforced with the "teach back" method in the preoperative period on postoperative mobilization in women who underwent gynecological oncology surgery.

DETAILED DESCRIPTION:
Mobilization; It is defined as "standing up, walking, being able to move and walking around, especially after the operation, when the patient stands up and walks around". Postoperative mobilization is a basic human need and one of the basic principles of nursing care. In the postoperative period, with the delay of mobilization, the patient's insulin resistance increases, muscle weakness and muscle mass loss occur, problems in pulmonary functions are experienced and the risk of thromboembolism increases. On the other hand, there is a significant relationship between increasing postoperative mobilization and postoperative recovery. It has been reported that day mobilization is significantly associated with successful surgical outcome and postoperative recovery (such as early return of bowel movements, shorter initiation of oral intake, shorter hospital stay).

Early mobilization after gynecological oncology surgeries is an important component of nursing care during the surgical process and one of the basic responsibilities of the surgical nurse. Within the scope of this responsibility, nurses should comprehensively evaluate patients physiologically and psychologically in the preoperative period, follow current evidence-based practices, and plan the nursing care process based on these practices in accordance with the clinical condition of the patient. It is reported that by following evidence-based practices in the treatment and care practices of patients in the postoperative period, the postoperative recovery process will be accelerated, the complications seen will be reduced, the hospital stay will be shortened, mortality and morbidity rates will be reduced, and patient satisfaction will be increased.

In this study, a systematic review and meta-analysis study was carried out to identify evidence-based interventions used to increase early postoperative mobilization and search PubMed, EBSCO (Medline, CINAHL), Web of Science, Cochrane, ClinicalTrials.gov and Turkey national databases (Dergipark, Turkey). Clinics, Turkmedline, and the National Thesis Center, Cochrane Library and TUBITAK Ulakbim databases were used in the last 20 years (01.01.2002-31.12.2022). Systematic reviews and meta-analyses published in Turkish and English are limited to observational studies, non-randomized and randomized controlled studies. Keywords were created according to the research question. MeSH (Medical Subject Headings) was used for English keywords, and Science Words of Turkey (SWT) was used to create Turkish equivalents of English keywords. The keywords used in the search were determined as "early ambulation" OR "early mobilization". The English keywords were determined as "Gynecologic Surgery" OR "Gynecological Surgery" OR "Gynecologic Surgical Procedure" OR "Gynecological Surgical Procedures" AND "Accelerated Ambulation" OR "Early Ambulation" OR "Early Mobilization". As a result of the screening, 6 studies that met the inclusion criteria and 2 interventions that were effective in increasing postoperative mobilization after gynecological oncology surgery were identified:

* Preoperative patient education,
* Exercise protocols. According to these results, it was decided to test the preoperative patient education in a randomized controlled experimental phase, considering the fact that this study is a doctoral thesis, the time limitation of the study, and the feasibility of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Having elective surgery
* Be conscious
* Having undergone gynecological oncological (vulva-vaginal cancer, ovarian cancer, cervical cancer, fallopian tube cancer, endometrial cancer) surgery
* Absence of mental and physical problems (such as Alzheimer's disease, dementia, orthopedic problems and limb amputation) that prevent early mobilization
* Having normal blood pressure and heart rate
* Being in ASA I, II and III classification
* Absence of abnormal findings at the incision site
* Have a phone number where you can be reached
* Permission of the physician (As the physician may recommend absolute bed rest to the patient in some cases in accordance with the clinical picture of the patients, the patient will not be included in the study in the presence of such a recommendation)

Exclusion Criteria:

* Being diagnosed with a neurological and/or psychiatric disorder
* Having a disability related to mobility
* Those with delirium in the postoperative period
* Patients with cardiac problems
* Patients with a history of diagnosed venous thrombosis
* Have had surgery in the last 1 month those who are pregnant
* Patients with a body temperature of 38.5 and above in the perioperative period
* Don't be intubated
* Lack of knowledge that he has been diagnosed with cancer (the case that the diagnosis is hidden from the patient)
* Using an assistive device for mobility
* Physician's written bed rest instruction
* Presence of abnormal finding in the surgical field
* Presence of a pacemaker
* Presence of respiratory diseases

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Patient mobility level | Postoperative day 1
  Assessed with Patient Mobility Scale. The scale is used to evaluate patient perceptions and objective observations regarding postoperative patient mobility. The scale questions are related to the severity of pain derived from the five-point likert scale, and for each item in the scale, the participants said "no pain" (1 point); "a mild pain" (2 points); "moderate pain" (3 points); They are asked to mark as "extreme pain" (4 points) and "the worst pain they can imagine" (5 points). The scores from all activities are added together to calculate the scores from the scale. The lowest score that can be obtained from the scale is 0, and the highest score is 120. A higher total score from the scale indicates increased pain and difficulty associated with activity.
Patient mobility level | Postoperative day 2
  Assessed with Patient Mobility Scale just as postoperative day 1. The lowest score that can be obtained from the scale is 0, and the highest score is 120. A higher total score from the scale indicates increased pain and difficulty associated with activity. (Repeated measure).
Patient mobility level | Postoperative day 3
  Assessed with Patient Mobility Scale just as postoperative day 1 and 2. The lowest score that can be obtained from the scale is 0, and the highest score is 120. A higher total score from the scale indicates increased pain and difficulty associated with activity. (Repeated measure).
Observer mobility level | Postoperative day 1.
  Assessed with Observer Mobility Scale. Observer Mobility Scale, During the performance of 4 activities (turning from side to side in the bed, sitting by the bed, standing up by the bed and walking in the patient room) after the surgical intervention, addiction was assessed. The state/degree of independence is scored between "1" and "5". The scores for the 4 activities are added together to calculate the scale score. The lowest and highest score that can be obtained from the scale is between 4-20. The increase in the score indicates that the mobility skills of the patients are insufficient, and the decrease in the score indicates that their ability to move after the surgical intervention is good/sufficient.
Observer mobility level | Postoperative day 2
  Assessed with Observer Mobility Scale just as postoperative day 1. The lowest and highest score that can be obtained from the scale is between 4-20. The increase in the score indicates that the mobility skills of the patients are insufficient, and the decrease in the score indicates that their ability to move after the surgical intervention is good/sufficient. (Repeated measure).
Observer mobility level | Postoperative day 3 just as postoperative day 1.
  Assessed with Observer Mobility Scale just as postoperative day 1. The lowest and highest score that can be obtained from the scale is between 4-20. The increase in the score indicates that the mobility skills of the patients are insufficient, and the decrease in the score indicates that their ability to move after the surgical intervention is good/sufficient. (Repeated measure).
The surgical recovery status after intervention | Postoperative day 3
  assessed with Postoperative Recovery Index Form. There are 5 sub-dimensions of the scale; psychological symptoms, physical activities, general symptoms, intestinal symptoms, and craving-desire symptoms. The scores of the items included in the sub-dimensions are summed, their arithmetic average is taken, and the sub-dimension score is determined. For the total score of scale; all 25 items are summed and the arithmetic average is taken. The total score that can be obtained from the index is reported as 25 (minimum) and 175 (maximum). The index can be applied any time between the 1st day and the 30th day after surgery. High scores from the index reflect more difficulty in post-operative recovery, while low scores indicate that recovery is easier after surgery.
The surgical recovery status after intervention | Postoperative day 15
  assessed with Postoperative Recovery Index Form just as postoperative day 3. The total score that can be obtained from the index is reported as 25 (minimum) and 175 (maximum). The index can be applied any time between the 1st day and the 30th day after surgery. High scores from the index reflect more difficulty in post-operative recovery, while low scores indicate that recovery is easier after surgery. (Repeated mesure).
Care satisfaciton | Postoperative third day
  assessed with Newcastle Nursing Care Satisfaction Scale. In this study, only the scale part of the scale will be used. The 19 items in the scale are 5-point likert-type and aim to describe the satisfaction of patients in various aspects of nursing care. In the scoring used to determine the degree of satisfaction; 1- I was never satisfied, 2- I was rarely satisfied, 3- I was satisfied, 4- I was very satisfied, 5- I was completely satisfied. The scale has no cut-off point. With the scale, the satisfaction of the patient in terms of nursing is evaluated as long as the patient stays in the patient's room. Score evaluation is made over 0-100 points by converting to 100 after the scores of all items in the scale are summed. It is reported that a total score of 100 indicates satisfaction with all aspects of nursing care.

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi Arslan, Principal Investigator — Aydın Adnan Menderes University, Faculty of Nursing, Surgical Nursing Department
Locations (1):
- Aydın Adnan Menderes University, Efeler, Aydın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: CSR
Time Frame: 12 months after publication
Access Criteria: Relevance to the topic of the study and approval of all-authors within 1 month of receiving the request.

REFERENCES:
- [Derived] Arslan E, Ozkan S. Effects of Preoperative Mobilization Education Using the Teach-Back Method on Patient Outcomes After Gynecological Surgery: A Randomized-Controlled Study. Nurs Health Sci. 2025 Jun;27(2):e70151. doi: 10.1111/nhs.70151. PMID 40442058